CLINICAL TRIAL: NCT02082678
Title: Ondansetron for Bipolar Disorder and Alcohol Use Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112013-075
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Alcohol Use Disorder; Dual Diagnosis
Keywords: Bipolar Disorder; BPD; Alcohol Use Disorder; Alcohol Abuse; Alcohol Dependence; Ondansetron; Cognition; Mood
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Active Comparator): Ondansetron will be given 0.5 mg twice a day (BID). The dose may be increased from 0.5 mg/BID to 1.0 mg/BID at week 4 for participants with less than 30% reduction in HAMD and/or alcohol use. An additional dose increase to 2.0 mg/BID and 4.0 mg/BID is allowed at weeks 8 and 10, respectively, for participants with less than a 50% reduction in HAMD scores and/or alcohol use.
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): Placebo will be given 0.5 mg/ BID. The dose may be increased from 0.5 mg/BID to 1.0 mg/BID at week 4 for participants with less than 30% reduction in HAMD and/or alcohol use. An additional dose increase to 2.0 mg/BID and 4.0 mg/BID is allowed at weeks 8 and 10, respectively, for participants with less than a 50% reduction in HAMD scores and/or alcohol use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Ondansetron is a serotonin receptor antagonist that is FDA-approved to treat nausea and vomiting caused by cancer therapy and surgery.
  Other Names: Zofran; Zuplenz
  Arms: Ondansetron
Drug: Placebo — Inactive ingredient matching the active medication in appearance
  Other Names: Sugar-pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if ondansetron, as an add-on therapy, is associated with reduced depressive symptoms and alcohol use in outpatients with bipolar disorder (BPD), cyclothymic disorder, schizoaffective disorder (bipolar type) and major depressive disorder (MDD) with mixed features. The investigators will also use blood samples to determine if the genotype for the serotonin transporter gene is associated with response to ondansetron.

DETAILED DESCRIPTION:
A total of 70 outpatients with alcohol use disorder and BPD, cyclothymic disorder, schizoaffective disorder (bipolar type), or MDD with mixed features will be enrolled in a 12-week, randomized, double-blind, parallel-group, placebo-controlled study of ondansetron. Participant will receive either ondansetron or a placebo for 12 weeks. He or she has an equal chance of receiving ondansetron or placebo.

Randomization will be stratified based on > 4 or ≤ 4 drinking days per week at start of the study. Ondansetron or placebo will be given at 0.5 milligrams twice a day for the first 4 weeks. At weeks 4, 8 and 10 the dose may be increased to 1.0, 2.0 or 4.0 milligrams twice a day, respectively, if significant reductions in depression and alcohol use are not observed and the participant is not experiencing any side effects. Blood will be drawn for routine laboratory analyses including a complete blood count (CBC), liver panel, and Carbohydrate-deficient Transferrin (CDT) at baseline and weeks 4, 8 and 12.

Each participant will return for weekly follow-up visits and repeat outcome measures. Pill counts will be conducted, and a list of current medications and doses will be recorded at each visit. Participants will be compensated at each appointment with a bus pass, gift cards, and a monetary incentive for compliance. Participants will be evaluated by both the research assistant (RA) and principal investigator (PI) at each visit.

The Hamilton Rating Scale for Depression (HAMD) and Timeline Followback (TLFB) will be given at each visit as the primary outcome measures. Cognitive assessments will be performed at baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18-70 years old with bipolar I, II, or Not Otherwise Specified (NOS) disorders, schizoaffective disorder (bipolar type), cyclothymic disorder, or major depressive disorder with mixed features
* Current diagnosis of alcohol use disorder (DSM V terminology) with onset ≤ age 25
* Alcohol use (by self-report) of at least 15 drinks in the 7 days prior to intake
* IF diagnosis of Bipolar I, II, or NOS Disorder: Current mood stabilizer therapy (lithium, anticonvulsant, atypical antipsychotic) with stable dose for at least 14 days prior to randomization
* IF diagnosis of Schizoaffective disorder (bipolar type): Current atypical antipsychotic therapy with stable dose for at least 14 days prior to randomization
* IF diagnosis of Major Depressive Disorder with mixed features: Current antidepressant therapy with stable dose for at least 14 days prior to randomization

Exclusion Criteria:

* Baseline Young Mania Rating Scale (YMRS) or Hamilton Rating Scale for Depression (HAMD) scores ≥ 35 to exclude those with very severe mood symptoms
* Evidence of clinically significant alcohol withdrawal symptoms defined as a CIWA-Ar (Clinical Institute Withdrawal Assessment of Alcohol Use-Revised) score of ≥ 10
* Therapy in past 14 days with naltrexone, acamprosate, disulfiram, or topiramate
* Vulnerable populations (e.g. pregnant, breastfeeding, incarcerated, cognitively impaired (e.g. dementia, mentally challenged))
* High risk of suicide defined as > 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded
* Intensive outpatient treatment (defined as ≥ 3 visits each week) for substance abuse (AA, NA meetings, or less intensive counseling at baseline will be allowed)
* Severe or life-threatening medical condition (e.g., hepatic cirrhosis) or laboratory or physical examination findings consistent with serious medical illness (e.g., dangerously abnormal electrolytes)
* AST (aspartate aminotransferase ) or ALT (alanine transaminase) > 3 times the upper limit of normal
* History of severe side effects or allergic reaction with prior ondansetron therapy (e.g. for vomiting) or use of medications with significant drug-drug interactions with ondansetron (phenytoin, carbamazepine, and rifampicin, apomorphine, tramadol)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron: Ondansetron will be given at the dose of 0.5 mg twice a day. The dose may be increased from 0.5 mg twice a day to 1.0 mg twice a day at week 4 for participants with less than 30% reduction in the Hamilton Depression Rating Scale (HAMD) and/or alcohol use based on Timeline Followback (TLFB) assessment of alcohol use. An additional dose increase to 2.0 mg twice a day and 4.0 mg twice a day is allowed at weeks 8 and 10, respectively, for participants with less than a 50% reduction in HAMD scores and/or TLFB.
- Placebo: Placebo that matches the active medication in appearance will be started at 0.5 mg capsule twice day. The dose may be increased from 0.5 mg twice day to 1.0 mg twice a day at week 4 for participants with less than 30% reduction in the Hamilton Depression Rating Scale (HAMD) and/or alcohol use per Timeline Followback (TLFB) assessment score. An additional dose increase to 2.0 mg twice a day and 4.0 mg twice a day is allowed at weeks 8 and 10, respectively, for participants with less than a 50% reduction in HAMD scores and/or alcohol use per TLFB.
Period: Overall Study
Arm/Group | Ondansetron | Placebo
Started | 35 | 35
Completed | 23 | 21
Not Completed | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Ondansetron: Ondansetron will be given 0.5 mg/ BID. The dose may be increased from 0.5 mg/BID to 1.0 mg/BID at week 4 for participants with less than 30% reduction in HAMD and/or alcohol use. An additional dose increase to 2.0 mg/BID and 4.0 mg/BID is allowed at weeks 8 and 10, respectively, for participants with less than a 50% reduction in HAMD scores and/or alcohol use.
  Ondansetron: Ondansetron is a serotonin receptor antagonist that is FDA-approved to treat nausea and vomiting caused by cancer therapy and surgery.
- Total: Total of all reporting groups
Arm/Group | Ondansetron | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 24 | 18 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 18 | 36
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.54 (8.60) | 43.29 (10.01) | 44.91429 (9.41128)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HAMD)
Description: The Hamilton Rating Scale for Depression (HAMD) is a 17-item observer-rated measure of depressive symptomatology. HAMD is scored between 0 and 4 points, with the total score ranging from 0 to 52. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression. The higher scores are associated with greater depressive symptom severity and poorer outcome.
Time Frame: Baseline and Week 12
Population: 11 participants from Ondansetron group and 13 from the Placebo group did not complete this study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 13.77 (5.39) | 14.23 (7.25)
  Week 12 | 8.52 (6.02) | 8.86 (5.77)

2. Primary Outcome: Number of Standard Drinks Per Assessment Period on Timeline Followback (TLFB)
Description: The Timeline Followback (TLFB) will be used to assess the change in the number of standard alcoholic drinks per week. The TLFB is interviewer-administered and asks participants to retrospectively estimate their alcohol use between each visit. The reported drinks are then converted to standard drinks based on the drink's alcohol by volume (ABV). The higher number is associated with more standard drinks and worse outcome. Values are corrected for the number of days covered in the assessment period.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: mean number of standard drinks per week
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 35 | 35
mean number of standard drinks per week
  Baseline | 4.06 (4.07) | 4.92 (4.09)
  Week 12 | 2.50 (3.73) | 2.92 (2.68)

3. Primary Outcome: Number of Heavy Drinking Days Per Assessment Period on Timeline Followback (TLFB)
Description: The Timeline Followback (TLFB) will be used to assess the change in the number of standard alcoholic drinks per week. The TLFB involves asking participants to retrospectively estimate their alcohol between each research visit. The reported drinks are then converted to heavy drinking days based on the drink's alcohol by volume (ABV) and participant's sex (male/female) - 5 drinks per day for males and 4 for females. Each day during which 4-5 drinks are consumed is counted as a heavy drinking day within a given assessment period. The reported values are corrected for days covered (divided by the number of days between each visit). The higher number is associated with more heavy drinking days and worse outcome.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: heavy drinking days (corrected)
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 35 | 35
heavy drinking days (corrected)
  Baseline | 0.34 (0.33) | 0.45 (0.37)
  Week 12 | 0.17 (0.28) | 0.20 (0.28)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were assessed by a weekly questionnaire at each appointment.
Arm/Group | Ondansetron | Placebo
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 10/35 | 4/35
Other Adverse Events (participants affected / at risk) | 7/35 | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron (N=35) | Placebo (N=35)
UTI (Infections and infestations) | 1 (1) | 0 (0)
Bacterial parasite in gut (Infections and infestations) | 1 (1) | 0 (0)
Leg swelling (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Detoxification (Social circumstances) | 1 (1) | 0 (0)
Suicide attempt (Social circumstances) | 1 (1) | 1 (1) — Overdose
Manic episode (Psychiatric disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Corneal ulcer (Infections and infestations) | 1 (1) | 0 (0)
Spinal disk degeneration (Nervous system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Suicide ideation (Social circumstances) | 1 (1) | 1 (1)
Prolonged QTc interval (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondansetron (N=35) | Placebo (N=35)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in finger and foot (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Sedation (General disorders) | 0 (0) | 1 (1)
Auditory hallucinations (Psychiatric disorders) | 0 (0) | 2 (2)
Swollen feet (General disorders) | 1 (1) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Suicidal ideation (Social circumstances) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02082678/Prot_SAP_000.pdf